CLINICAL TRIAL: NCT04458272
Title: A Phase II Study of DS-1001b in Patients With Chemotherapy- and Radiotherapy-naive IDH1 Mutated WHO Grade II Glioma
Brief Title: A Study of DS-1001b in Patients With Chemotherapy- and Radiotherapy-Naive IDH1 Mutated WHO Grade II Glioma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS1001-A-J201; 205339 (Other: JapicCTI)
Record Dates: First submitted 2020-06-29; First posted 2020-07-07 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: WHO Grade II Glioma
Keywords: DS-1001; IDH1; Glioma; IDH-mutant glioma; WHO grade II glioma; Low-grade glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DS-1001b (Experimental)
  Interventions: Drug: DS-1001b

INTERVENTIONS:
Drug: DS-1001b — 250 mg, twice daily, continuous oral administration

SUMMARY:
This Phase 2 study is conducted to assess the efficacy and safety of DS-1001b in patients with chemotherapy- and radiotherapy-naive IDH1 mutated WHO grade II glioma.

ELIGIBILITY:
Inclusion Criteria:

* Has a histopathologically documented IDH1 mutated WHO grade II glioma according to the 2016 WHO classification.
* Has confirmed IDH1 mutation at the R132 locus by testing at the central laboratory conducted during the screening period.
* Has no prior anticancer treatment (including chemotherapy and radiotherapy) for glioma except craniotomy or biopsy.
* Has at least 1 measurable and non-enhancing lesion.
* Has an interval of at least 90 days from the latest surgery.
* Has no sign of malignant transformation including the appearance of enhancing lesions and/or rapid growth of non-enhancing lesions.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 1.

Exclusion Criteria:

* Has had a histopathological diagnosis of WHO grade III or IV glioma.
* Has had a contrast enhancing lesion on brain MRI.
* Has received a prior treatment with any mutant IDH1 inhibitor.
* Has received other investigational products within 28 days before the start of the study drug treatment.
* Has an active infection requiring systemic treatment.
* Has multiple primary malignancies.
* Has a history of clinically significant cardiac disease.
* Is a pregnant or lactating woman.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) assessed by Independent Efficacy Review Committee | Up to 24 months
Number of participants with treatment-emergent adverse events (TEAEs) during the study | Up to 24 months

SECONDARY OUTCOMES:
Clinical benefit rate | Through the end of the study (up to approximately 6 years)
Percentage change in tumor volume | Through the end of the study (up to approximately 6 years)
Time to response | Through the end of the study (up to approximately 6 years)
Duration of response | Through the end of the study (up to approximately 6 years)
Time to treatment failure | Through the end of the study (up to approximately 6 years)
Progression-free survival | Through the end of the study (up to approximately 6 years)
Overall survival | Through the end of the study (up to approximately 6 years)
Area under the concentration curve (AUC) for DS-1001a | Cycle 1 Day 1 to Cycle 13 Day 1 (each cycle is 28 days)
Maximum plasma concentration (Cmax) for DS-1001a | Cycle 1 Day 1 to Cycle 13 Day 1 (each cycle is 28 days)
Time to maximum plasma concentration (Tmax) for DS-1001a | Cycle 1 Day 1 to Cycle 13 Day 1 (each cycle is 28 days)
Change from baseline in 2-hydroxyglutarate (2-HG) concentration in patient specimens after treatment with DS-1001b | Through the end of the study (up to approximately 6 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (11):
- Japan (11):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Hiroshima University Hospital, Hiroshima
  - Kumamoto University Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - National Hospital Organization Osaka National Hospital, Osaka
  - Kyorin University Hospital, Tokyo
  - National Cancer Center Hospital, Tokyo
  - Tokyo Women's Medical University Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Arakawa Y, Saito R, Kanemura Y, Mishima K, Koriyama S, Narita Y, Kumabe T, Motomura K, Sugiyama K, Yamasaki F, Mukasa A, Kanamori M, Kuga D, Nagane M, Kakurai Y, Isobe K, Nakamura H. Phase II study of safusidenib erbumine in patients with chemotherapy- and radiotherapy-naive isocitrate dehydrogenase 1-mutated WHO grade 2 gliomas. Neuro Oncol. 2025 Nov 8:noaf258. doi: 10.1093/neuonc/noaf258. Online ahead of print. PMID 41206766
- [Derived] Natsume A, Arakawa Y, Narita Y, Sugiyama K, Hata N, Muragaki Y, Shinojima N, Kumabe T, Saito R, Motomura K, Mineharu Y, Miyakita Y, Yamasaki F, Matsushita Y, Ichimura K, Ito K, Tachibana M, Kakurai Y, Okamoto N, Asahi T, Nishijima S, Yamaguchi T, Tsubouchi H, Nakamura H, Nishikawa R. The first-in-human phase I study of a brain-penetrant mutant IDH1 inhibitor DS-1001 in patients with recurrent or progressive IDH1-mutant gliomas. Neuro Oncol. 2023 Feb 14;25(2):326-336. doi: 10.1093/neuonc/noac155. PMID 35722822